CLINICAL TRIAL: NCT02780219
Title: The Effects of Acute Resistance Exercise on Protein and Amino Acid Metabolism in Chronic Obstructive Pulmonary Disease
Brief Title: Chronic Obstructive Pulmonary Disorder and Acute Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Non-Randomized | Model: Single Group | Purpose: Supportive Care
Other Study IDs: 2015-0768
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy (Experimental): screening visit: body weight and composition by DXA, height, and vital signs will be assessed.
  study day(s): may include combinations of stable isotope infusions with blood draws, acute exercise, cognition testing
  Interventions: Other: stable amino acid infusion; Other: acute exercise with amino acid infusion; Other: 24-hour post exercise amino acid infusion
- Chronic Obstructive Pulmonary Disorder (Experimental): screening visit: body weight and composition by DXA, height, and vital signs will be assessed.
  study day(s): may include combinations of stable isotope infusions with blood draws, acute exercise, cognition testing
  Interventions: Other: stable amino acid infusion; Other: acute exercise with amino acid infusion; Other: 24-hour post exercise amino acid infusion

INTERVENTIONS:
Other: stable amino acid infusion — stable isotopes Such as L-[ring-13C6]-Phenylalanine, L-[ring-D4]Tyrosine, L-[Methyl-D3]Tau-Methylhistidine, trans-[2,5,5-D3]4-Hydroxy-L-proline, L-[Guanido-15N2]-Arginine, L-[4,4,5,5-D4-5-13C]Citruline, L-13C5 -Ornithine, L-15N2-Glutamine, L-[1,2-13C2]Glutamic Acid, 1-13C-Glycine, L-15N3-Histidine, L-13C6-Leucine, L-[methyl-D3]Methionine, α-1-13C-ketoisocaproic acid, L-1-13C-Methionine, DL-[3,3,4,4-D4]Homocysteine, L-[1,2-13C2]Taurine, L-(Indole-D5)Tryptophan, 13C-Urea, L-1-13C-Isoleucine, L-13C5-Valine, α-[Dimethyl-13C2]ketoisovaleric acid, 2-keto-3-methyl-13C6-pentanoate, 3-hydroxy-[3,4-methyl-13C3]isovaleric acid, 13C3-glycerol is given IV simultaneously
Other: acute exercise with amino acid infusion — resistance exercise of each limb (i.e., leg (right/left); arm (right/left) on an isokinetic exercise machine allowing control of velocity, force, etc. with stable isotopes such as L-[ring-13C6]-Phenylalanine, L-[ring-D4]Tyrosine, L-[Methyl-D3]Tau-Methylhistidine, trans-[2,5,5-D3]4-Hydroxy-L-proline, L-[Guanido-15N2]-Arginine, L-[4,4,5,5-D4-5-13C]Citruline, L-13C5 -Ornithine, L-15N2-Glutamine, L-[1,2-13C2]Glutamic Acid, 1-13C-Glycine, L-15N3-Histidine, L-13C6-Leucine, L-[methyl-D3]Methionine, α-1-13C-ketoisocaproic acid, L-1-13C-Methionine, DL-[3,3,4,4-D4]Homocysteine, L-[1,2-13C2]Taurine, L-(Indole-D5)Tryptophan, 13C-Urea, L-1-13C-Isoleucine, L-13C5-Valine, α-[Dimethyl-13C2]ketoisovaleric acid, 2-keto-3-methyl-13C6-pentanoate, 3-hydroxy-[3,4-methyl-13C3]isovaleric acid, 13C3-glycerol is given IV simultaneously
Other: 24-hour post exercise amino acid infusion — stable isotopes such as L-[ring-13C6]-Phenylalanine, L-[ring-D4]Tyrosine, L-[Methyl-D3]Tau-Methylhistidine, trans-[2,5,5-D3]4-Hydroxy-L-proline, L-[Guanido-15N2]-Arginine, L-[4,4,5,5-D4-5-13C]Citruline, L-13C5 -Ornithine, L-15N2-Glutamine, L-[1,2-13C2]Glutamic Acid, 1-13C-Glycine, L-15N3-Histidine, L-13C6-Leucine, L-[methyl-D3]Methionine, α-1-13C-ketoisocaproic acid, L-1-13C-Methionine, DL-[3,3,4,4-D4]Homocysteine, L-[1,2-13C2]Taurine, L-(Indole-D5)Tryptophan, 13C-Urea, L-1-13C-Isoleucine, L-13C5-Valine, α-[Dimethyl-13C2]ketoisovaleric acid, 2-keto-3-methyl-13C6-pentanoate, 3-hydroxy-[3,4-methyl-13C3]isovaleric acid, 13C3-glycerol is given IV simultaneously

SUMMARY:
For this study a resistance bout will be performed in order to promote the robust response of protein synthesis. Type II muscle fibers often exhibit more atrophy than type I fibers in COPD subjects therefore specifically targeting them in an exercise protocol could have more beneficial outcome for these individuals.

DETAILED DESCRIPTION:
In this study, the following hypothesis will be tested: A bout of resistance exercise will affect the acute and 24h response in whole-body protein and amino acid metabolism and cognitive function as compared to baseline values in COPD patients and healthy subjects. To do this, subjects will complete a baseline visit in which they receive stable amino acid tracers. The next day they will complete a one-time resistance exercise with an immediate measurement of the amino acid tracers, and return 24 hours after exercise to repeat amino acid tracer measurements. This project will provide important clinical information on the whole body protein and amino acid metabolic response to acute resistance exercise in elderly subjects with COPD, as well as, the exercise induced changes in physical and cognitive function, and absolute muscular strength capacity in this population. In this way, this study will provide preliminary data for the development of standardized, repeatable resistance exercise protocols that will stop the process of ongoing muscle loss and improve metabolism and function in COPD subjects.

ELIGIBILITY:
Inclusion criteria COPD subjects:

* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lie in supine or elevated position for 4 hours
* Diagnosis of moderate to very severe chronic airflow limitation and compliant to the following criteria: FEV1 < 70% of reference FEV1
* Clinically stable condition and not suffering from a respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding year) at least 4 weeks prior to the first test day
* Shortness of breath on exertion
* Willingness and ability to comply with the protocol

Inclusion criteria healthy subjects:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lay in supine or elevated position for 4 hours
* No diagnosis of COPD
* Willingness and ability to comply with the protocol

Exclusion Criteria all subjects:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (healthy subjects only)
* Established diagnosis of malignancy
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Body mass index >40 kg/m2 (healthy subjects only)
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* Use of protein or amino acid containing nutritional supplements within 5 days of first study day
* Previous injury that could interfere with participation in resistance exercise protocol
* Use of short course of oral corticosteroids within 4 weeks preceding first study day
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* (Possible) pregnancy
* Already enrolled in another clinical trial and that clinical trial interferes with participating in this study

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Change in net whole-body protein synthesis | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
  Change in whole-body protein synthesis rate

SECONDARY OUTCOMES:
glutamate related metabolism | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
tryptophan related metabolism | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
arginine related metabolism | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
leucine related metabolism | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
taurine related metabolism | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
Body Composition | 15 minutes on screening or study day 1
  Body composition as measured by Dual-Energy X-ray Absorptiometry
changes in skeletal muscle fatigue | on study day 1 and change from day 2 and day 3
  kin-com 1-leg test
Group differences in state of mood as measured by the Hospital Anxiety and Depression Scale (HADS) | 1 day
  a fourteen item self-assessment scale. Seven of the items related to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression.
Group differences in attention and executive functions as measured by Stroop Color-Word Test (SCWT) | on study day 1 and change from day 2 and day 3
  a word page with words printed in black ink, a color page with blocks printed in color, and a color-word page where the color and the word do not match. The examinee reads the words or names the ink colors as quickly as possible within a time limit. Measures selective attention and inhibitory control. The total time in seconds was reported for each trial.
Group differences in learning and memory as measured by Digit Span | on study day 1 and change from day 2 and day 3
  recall of numbers in the same order (Digit Forward) and in reverse order (Digit Backward). Measures auditory attention and verbal working memory.
Group differences in attention and executive functions as measured by Digit Symbol Modalities Test | on study day 1 and change from day 2 and day 3
  Using a legend with nine symbols that correspond to nine different numbers, the examinee is asked to fill in as many blank squares as possible by copying the corresponding number in each box, indexed by a symbol within a 90 sec time limit.
Group differences in activity as measured by Physical Activity Scale for the Elderly (PASE) | study day 1
  This questionnaire is intended for use in an elderly population and focuses on 3 types of activities: leisure time activities, household activities and work-related activities.
24 hour diet recall | study day 1
  The subject is asked to recall in detail all the food and drink consumed during the 24 hours prior to the test day.
appetite questionnaire | study day 1
  The subject is asked to rate various aspects of their appetite as relates to overall health

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University-CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sontam T, Deutz NEP, Cruthirds CL, Mbilinyi R, Ruebush LE, Ten Have GA, Thaden JJ, Engelen MPKJ. Prolonged disturbances in citrulline metabolism following resistance exercise in COPD. Clin Nutr. 2025 Jun;49:21-32. doi: 10.1016/j.clnu.2025.03.021. Epub 2025 Apr 8. PMID 40233541
- [Derived] Mbilinyi RH, Deutz NEP, Cruthirds CL, Ruebush LE, Sontam T, Ten Have GAM, Thaden JJ, Engelen MPKJ. Prolonged increase in glutamate whole body and intracellular production in older adults with COPD and healthy controls post-resistance exercise. Metabolism. 2025 Jul;168:156185. doi: 10.1016/j.metabol.2025.156185. Epub 2025 Mar 18. PMID 40113079
- [Derived] Deutz LN, Wierzchowska-McNew RA, Deutz NE, Engelen MP. Reduced plasma glycine concentration in healthy and chronically diseased older adults: a marker of visceral adiposity? Am J Clin Nutr. 2024 Jun;119(6):1455-1464. doi: 10.1016/j.ajcnut.2024.04.008. Epub 2024 Apr 12. PMID 38616018
- [Derived] Engelen MPKJ, Kirschner SK, Coyle KS, Argyelan D, Neal G, Dasarathy S, Deutz NEP. Sex related differences in muscle health and metabolism in chronic obstructive pulmonary disease. Clin Nutr. 2023 Sep;42(9):1737-1746. doi: 10.1016/j.clnu.2023.06.031. Epub 2023 Jul 26. PMID 37542951
- [Derived] Wierzchowska-McNew RA, Engelen MPKJ, Thaden JJ, Ten Have GAM, Deutz NEP. Obesity- and sex-related metabolism of arginine and nitric oxide in adults. Am J Clin Nutr. 2022 Dec 19;116(6):1610-1620. doi: 10.1093/ajcn/nqac277. PMID 36166849